CLINICAL TRIAL: NCT07111221
Title: A Prospective, Randomized Study Evaluating the Effectiveness of Portal Hypertension Modulation in the Preoperative Period in Patients at Increased Risk of Massive Blood Loss During Liver Transplantation.
Brief Title: Portal Inflow Modulation Prior to Liver Transplantation in Patients With Increased Risk of Intraoperative Blood Loss
Acronym: PIMLivT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ABM32
Record Dates: First submitted 2025-07-21; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-06

CONDITIONS: Liver Cirrhosis; Clinically Significant Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-selective beta blockers (Active Comparator): Non-selective beta blockers for treatment of portal hypertension
  Interventions: Drug: Non-selective beta-blockers
- Non-selective beta blockers + TIPS (Experimental): Non-selective beta blockers and TIPS for treatment of portal hypertension
  Interventions: Procedure: Transjugular Intrahepatic Portosystemic Shunt; Drug: Non-selective beta-blockers

INTERVENTIONS:
Procedure: Transjugular Intrahepatic Portosystemic Shunt — Transjugular Intrahepatic Portosystemic Shunt performed prior to liver transplantation in patients with increased risk of intraoperative blood loss
  Other Names: TIPS
  Arms: Non-selective beta blockers + TIPS
Drug: Non-selective beta-blockers — Non-selective beta-blockers for lowering portal hypertension
  Other Names: NSBBs

SUMMARY:
Liver transplantation is a procedure associated with an exceptionally high risk of blood loss. Liver failure, which is the most common indication for transplantation, not only leads to coagulation disorders but also to the development of portal hypertension. As a result, collateral circulation forms within the abdominal venous system, significantly increasing the risk of massive intraoperative blood loss. The number of intraoperatively transfused units of red blood cell concentrate is one of the main predictors of serious complications and postoperative mortality.

Patients with portal hypertension awaiting liver transplantation should be treated with non-selective β-blockers, which reduce pressure in the portal system. This is primarily justified by the need to prevent esophageal variceal bleeding, one of the most common causes of decompensation in chronic liver failure and a potential cause of death while awaiting liver transplantation.

According to the Baveno VII guidelines, if bleeding recurs despite the use of non-selective β-blockers, a transjugular intrahepatic portosystemic shunt (TIPS) should be considered. Significant reduction of portal pressure is observed in up to 50% of patients treated with propranolol and up to 75% with carvedilol. TIPS effectively prevents bleeding caused by portal hypertension.

However, recommendations for pre-transplant management of portal hypertension do not address the reduction of blood loss risk during liver transplantation. Previous studies evaluating the use of TIPS before transplantation primarily confirmed its safety and showed no significant increase in intraoperative risk. One analysis even suggested using TIPS in all patients with portal hypertension awaiting liver transplantation. Although some studies have addressed the issue of blood loss during transplantation, they were observational and retrospective, without distinguishing patients at particularly high risk of massive blood loss. So far, the effectiveness of TIPS in reducing blood loss during liver transplantation has not been confirmed-nor have studies reliably excluded such potential.

The objective of the study is to directly compare the effectiveness of two different methods of modulating portal hypertension in the context of the risk of massive blood loss during liver transplantation.

We hypothesize that the superior effectiveness of TIPS in significantly reducing portal hypertension may lead to a significant decrease in blood loss and the need for transfusion of blood products in patients at high risk of massive blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Qualification for elective liver transplantation from a deceased donor
* Age ≥18 years
* BMI between 18.5 kg/m² and 30 kg/m²
* Informed consent to participate in the study
* Clinically significant portal hypertension
* At least 1 of the following risk factors for massive blood loss:
* Re-transplantation
* Previous surgery in the upper abdomen
* History of esophageal variceal bleeding
* History of spontaneous bacterial peritonitis
* Planned thrombectomy during liver transplantation

Exclusion Criteria:

* Heart failure (EF <50%)
* Severe right ventricular failure
* Severe pulmonary hypertension
* Systemic infection
* Portal vein thrombosis (Yerdel >1)
* Severe coagulopathy (INR >5)
* Thrombocytopenia <20,000/ml
* Severe or uncontrolled encephalopathy (ammonia concentration >100 μmol/l)
* Contraindication to TIPS
* Contraindication to therapy with non-selective beta-blockers
* Pregnancy
* Lack of informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of red blood cell units transfused during liver transplantation. | Intraoperative

SECONDARY OUTCOMES:
Portal vein blood flow | Intraoperative
  Blood flow velocity in the portal vein during liver transplantation
Intraoperative blood loss | Intraoperative
  Blood loss during liver transplantation [ml]
Operation time | Intraoperative
  Time of surgery [min]
Postoperative complications | Up to 90 days
  CCI index and the percentage of complications ≥ grade 3 according to the Clavien-Dindo classification after liver transplantation
Time of hospitalisation | Up to 90 days
  Postoperative hospitalisation [days]
Variceal bleeding | Preoperative
  Esophageal variceal bleeding before transplantation
Overall survival | Up to 90 days
  Survival from the time of qualification for liver transplantation and up to 90 days after liver transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Centre of the Medical University of Warsaw, Warsaw, Poland